CLINICAL TRIAL: NCT03881930
Title: Balance REhabilitation With Modified Visual Input in Patients With acQuired Chronic Demyelinating Neuropathy and PROprioceptive Disorders
Brief Title: Balance Rehabilitation With Modified Visual Input in Patients With Neuropathy
Acronym: REQ-PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K170911J
Record Dates: First submitted 2019-01-25; First posted 2019-03-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Neuropathy; Ataxia; Proprioceptive Disorders; Balance; Distorted
Keywords: Peripheral neuropathy; Balance; Proprioceptive Disorders; Visual dependence; Rehabilitation; Physical Therapy
MeSH Terms: conditions — Ataxia; Somatosensory Disorders; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Observe in patients with chronic acquired demyelinating neuropathy, the effects on balance of a rehabilitation with modified visual input (deceived visual input, or visual deprivation); compared to an identical rehabilitation of balance performed with the non-modified visual input.
Who Masked: Outcomes Assessor
Masking Description: Evaluations are carried out outside the rehabilitation programme, by blind evaluators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Balance rehabilitation with modified visual input:
  In experimental group, patients with chronic acquired demyelinating neuropathy will benefit from 20 rehabilitation sessions with a Physical Therapist and 3 assessments.
  They will perform balance training with modified visual input.
  Interventions: Other: Balance rehabilitation with modified visual input
- control group (Active Comparator): Balance rehabilitation with no modified visual input:
  In control group, patients with chronic acquired demyelinating neuropathy will benefit from 20 rehabilitation sessions with a Physical Therapist and 3 assessments.
  They will perform balance training with no modified visual input.
  Interventions: Other: Balance rehabilitation with no modified visual input

INTERVENTIONS:
Other: Balance rehabilitation with modified visual input — Patients will perform the exercises alternatively: while keeping their eyes closed or their vision will be obstructed by a opaque mask or disturbed by moving luminous dots projected on the environment in a dark room without any visual reference cues.
  Arms: Experimental group
Other: Balance rehabilitation with no modified visual input — Patients will perform the exercises while keeping their eyes openned
  Arms: control group

SUMMARY:
This research focuses on the effects of rehabilitation on balance, in patients with acquired chronic demyelinating neuropathy. Rehabilitation will be performed with or without vision.

It is planned to include 40 subjects consulting for walking instability related to sensitivity disorders.

This multicenter study will take place in Paris's area. Each participant will benefit from 20 rehabilitation sessions with a Physical Therapist and 3 assessments.

Thanks to randomization, patient will be allocated in one of the 2 following groups:

* Control group, Patients will benefit from balance rehabilitation with open eyes.
* Experimental group, they will perform the same exercises while keeping their eyes closed or their vision will be obstructed by a mask or disturbed by moving luminous dots projected on the environment in darkness.

DETAILED DESCRIPTION:
Patients with chronic acquired demyelinating neuropathy may be referred for instability or falls when walking. Some of them have complaints of dysesthesia, paresthesia. The majority of these patients, due to the involvement of large sensory fibres, have deep and superficial sensitivity disorders (hypoesthesia or anaesthesia), which explain proprioceptive ataxia and balance disorders.

In a given situation, an individual maintains his or her balance thanks to sensory information, among which he or she may have to choose the most appropriate one for the context. A good balance control depends on the ability to select the best information, but many subjects do not have, or have lost, this ability, giving too systematically priority to the same sensory input. This is what is called sensory preferences or sensory profiles that differ from one subject to another. The most common behaviour is visual dependence.

This tendency to visual dependence has been described in different pathological situations, especially after a stroke. Research has shown that specific rehabilitation in visual deprivation can reduce visual dependence and improve balance and walking autonomy in stroke patients.

The investigators have shown in previous work that patients with acquired chronic demyelinating neuropathy have ataxic symptomatology with a visual dependence behavior, while a good sensitivity to vibration stimulation of proprioceptive pathways persists. The proprioceptive potential still present seems to be under-used.

Rehabilitation of patients with peripheral neuropathy involves many techniques, such as muscle strengthening, vibration, virtual reality, Tai chi, electrical stimulation, etc. However, some techniques, such as the use of virtual reality or visual biofeedback, tend to increase the use of the visual input, which could be detrimental to other inputs. The specific approach to balance disorders in these patients through manipulation of the visual input has, to our knowledge, not been studied. This is the objective of the study.

The main hypothesis of this research is that rehabilitation with modified visual input can, by reducing visual dependence, strengthen the proprioceptive input that still appears to be available in these patients with acquired chronic demyelinating neuropathy, despite deficits already present, and thus improve balance and walking ability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic demyelinating acquired neuropathy
* Age ≥ 18 years.
* Patients able to walk 20 meters without human assistance at least indoors with or without technical assistance.
* Patients with complaints such as discomfort, walking instability related to sensitivity disorders.
* Patients being clinically stable for at least 2 months, regardless of ongoing treatments.
* Patients who have provided consent.

Exclusion Criteria:

* Patients unable to walk 20 metres without technical and human assistance indoors.
* Patients with an ongoing hospitalization.
* Patients already included and participating in another intervention study.
* Patients with ongoing balance rehabilitation and continued during the REQ-PRO program in another rehabilitation centre or practice.
* Patients with ongoing acute treatment (related to polyneuropathy) started less than 2 months ago or stopped less than 2 months ago.
* Patients with scheduled surgery during the period of the patient's participation in the protocol, preventing the successful completion of the rehabilitation program and participation in assessments.
* Patients with recent surgery, in particular lower limb prosthesis (less than 1 year old) or equipment contraindicated for planned exercises such as standing kneeling positions.
* Patients with skin wounds on the foot that contraindicate rehabilitation.
* Patients with balance disorders of vestibular origin or central neurological pathology.
* Patients with a visual disability.
* Patients with a hearing impairment that prevents the patient from hearing and understanding instructions during the rehabilitation program or assessments.
* Patients with an inability to speak or understand the French language.
* Patients with cognitive or language impairments that prevent understanding of the protocol.
* Patients with a residence outside of the Paris Region (Ile de France).
* Patients with a known pregnancy.
* Patients not affiliated to a social security system (beneficiary or having a right), deprived of their right, under guardianship, curatorship, prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
U-turn time of realization, in seconds, realized at a comfortable speed measured with accelerometers just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session
  Evaluate balance during walking with a U-turn realized with eyes open at a comfortable speed by the time of realization, in seconds, of the U-turn, measured with accelerometers between 2 to 8 days after 20th and last rehabilitation session.

SECONDARY OUTCOMES:
U-turn time of realization, in seconds, realized at comfortable speed, measured with accelerometers 2 months after the end of the rehabilitation program. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn with eyes open realized at comfortable speed, by the time of realization, in seconds, of the U-turn measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
U-turn time of realization, in seconds, realized at fast speed, measured with accelerometers just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn with eyes open realized at fast speed, by the time of realization, in seconds, of the U-turn measured with accelerometers between 2 to 8 days after the 20th and last rehabilitation session
U-turn time of realization, in seconds, realized at fast speed, measured with accelerometers 2 months after the end of the rehabilitation program. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn with eyes open realized at fast speed, by the time of realization, in seconds, of the U-turn measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
Number of external steps of the U-turn realized at a comfortable speed, measured with accelerometers just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at comfortable speed by the number of external steps of the U-turn measured with accelerometers between 2 to 8 days after the 20th and last rehabilitation session.
Number of external steps of the U-turn realized at a comfortable speed, measured with accelerometers 2 months after the end of the rehabilitation program. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at a comfortable speed by the number of external steps of the U-turn measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
Number of external steps of the U-turn realized at fast speed, measured with accelerometers just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at fast speed by the number of external steps of the U-turn measured with accelerometers between 2 to 8 days after the 20th and last rehabilitation session.
Number of external steps of the U-turn realized at fast speed, measured with accelerometers 2 months after the end of the rehabilitation program. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at fast speed by the number of external steps of the U-turn measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
The double stance phase time, walking 20 meters, realized at a comfortable speed, measured with accelerometers just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at comfortable speed by the double stance phase in %, to walk 20 meters, measured with accelerometers between 2 to 8 days after the 20th and last rehabilitation session.
The double stance phase, walking 20 meters, realized at a comfortable speed, measured with accelerometers 2 months after the end of the rehabilitation program. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at a comfortable speed by the double stance phase in %, to walk 20 meters, measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
The double stance phase, walking 20 meters during walking with a U-turn, realized at fast speed, measured with accelerometers just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at fast speed by the double stance phase in %, to walk 20 meters, measured with accelerometers between 2 to 8 days after the 20th and last rehabilitation session.
The double stance phase, walking 20 meters, realized at fast speed, measured with accelerometers 2 months after the end of the rehabilitation program. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at fast speed by the double stance phase in %, to walk 20 meters, measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
Global amount of movement during walking with a U-turn realized at a comfortable speed, measured with accelerometers just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at comfortable speed by global amount of movement (related to oscillations and abruptness of the gesture) measured with accelerometers between 2 to 8 days after the 20th and last rehabilitation session.
Global amount of movement during walking with a U-turn, realized at a comfortable speed, measured with accelerometers 2 months after the end of the rehabilitation program. | between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at a comfortable speed by global amount of movement (related to oscillations and abruptness of the gesture), measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
Global amount of movement during walking with a U-turn realized at fast speed, measured with accelerometers just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at fast speed by the global amount of movement (related to oscillations and abruptness of the gesture), measured with accelerometers between 2 to 8 days after the 20th and last rehabilitation session.
Global amount of movement during walking with a U-turn realized at fast speed, measured with accelerometers 2 months after the end of the rehabilitation program. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance during walking with a U-turn realized with eyes open at fast speed by global amount of movement (related to oscillations and abruptness of the gesture), measured with accelerometers between 60 to 70 days after the 20th and last rehabilitation session.
Time in seconds, to walk 10 meters, realized with open eyes at a comfortable speed just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate the balance by the Time in seconds, to walk 10 meters, realized with open eyes at a comfortable speed between 2 to 8 days after the 20th and last rehabilitation session.
Time in seconds, to walk 10 meters, realized with open eyes at a comfortable speed 2 months after the end of the rehabilitation. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate the balance by the Time in seconds, to walk 10 meters, realized with open eyes at a comfortable speed between 60 to 70 days after the 20th and last rehabilitation session.
The number of steps, to walk 10 meters with open eyes at a comfortable speed just after the end of the rehabilitation | Between 2 to 8 days after the 20th and last rehabilitation session
  Evaluate the balance by the the number of steps, to walk 10 meters with open eyes at a comfortable speed between 2 to 8 days after the 20th and last rehabilitation session
The number of steps, to walk 10 meters with open eyes at a comfortable speed 2 months after the end of the rehabilitation | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate the balance by the the number of steps, to walk 10 meters with open eyes at a comfortable speed between 60 to 70 days after the 20th and last rehabilitation session
The Goggle Task performed just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session
  Evaluate the balance by the Goggle Task, the ratio: time in seconds, to walk 10 meters, in visual deprivation at comfortable speed / time in seconds, to walk 10 meters, eyes open at comfortable speed just after the end of the rehabilitation program.
The Goggle Task performed 2 months after the end of the rehabilitation | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate the balance by the Goggle Task, the ratio: time in seconds, to walk 10 meters, in visual deprivation at comfortable speed / time in seconds, to walk 10 meters, eyes open at comfortable speed between 60 to 70 days after the 20th and last rehabilitation session
The times, in seconds, of descent and ascent of a staircase floor, realized just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate balance by the times, in seconds, of descent and ascent of a staircase floor, realized with open eyes between 2 to 8 days after the 20th and last rehabilitation session.
The times, in seconds, of descent and ascent of a staircase floor, realized 2 months after the end of the rehabilitation | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance by the times, in seconds, of descent and ascent of a staircase floor, realized with open eyes between 60 to 70 days after the 20th and last rehabilitation session
Romberg quotient collected just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session
  Evaluate balance by the Romberg quotient collected during a static stabilometry test between 2 to 8 days after the 20th and last rehabilitation session.
Romberg quotient collected 2 months after the end of the rehabilitation | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate balance by the Romberg quotient collected during a static stabilometry test between 60 to 70 days after the 20th and last rehabilitation session.
Sensory preference realized just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session
  Determine the sensory profile of the patient by the sensory preference score after visual and proprioceptive stimuli between 2 to 8 days after the 20th and last rehabilitation session
Sensory preference realized 2 months after from the end of the rehabilitation | between 60 to 70 days after the 20th and last rehabilitation session
  Determine the sensory profile of the patient by the sensory preference score after visual and proprioceptive stimuli between 60 to 70 days after the 20th and last rehabilitation session
Monofilament test 10 g just after the end of the rehabilitation program. | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate the superficial sensitivity to tact on the sole of the foot by the monofilament test 10 g (Semmes-Weinstein 5.07) between 2 to 8 days after the 20th and last rehabilitation session.
Monofilament test 10 g, 2 months after the end of the rehabilitation. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate the superficial sensitivity to tact on the sole of the foot by the monofilament test 10 g (Semmes-Weinstein 5.07) between 60 to 70 days after the 20th and last rehabilitation session.
Score of kinesthetic sensitivity in the lower limbs just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session
  Evaluate sensitivity by a score of kinesthetic sensitivity in the lower limbs between 2 to 8 days
Score of kinesthetic sensitivity in the lower limbs, 2 months after the end of the rehabilitation. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate sensitivity by a score of kinesthetic sensitivity in the lower limbs between 60 to 70 days
Merkies palatal score in the lower limbs just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session
  Evaluate sensitivity by the Merkies palatal score in the lower limbs between 2 to 8 days after the 20th and last rehabilitation session.
Merkies palatal score in the lower limbs 2 months after the end of the rehabilitation | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate sensitivity by the Merkies palatal score in the lower limbs between 60 to 70 days after the 20th and last rehabilitation session
Simplified version of the "Activities-specific Balance Confidence scale just after the end of the rehabilitation program | Between 2 to 8 days after the 20th and last rehabilitation session.
  Evaluate the person's confidence in his or her balance, in the activities of daily living Simplified version of the "Activities-specific Balance Confidence scale between 2 to 8 days:the 20th and last rehabilitation session.
  Questionnaire made of 15 statements to assess the person's degree of confidence in his or her balance associated with activities of daily life in both the home environment and in the community environment. The questionnaire is part of this research administered by the evaluator.
  Add the scores obtained to the 15 items to obtain an overall score out of 45. The score is converted to a pourcentage.
Simplified version of the "Activities-specific Balance Confidence scale 2 months after the end of the rehabilitation. | Between 60 to 70 days after the 20th and last rehabilitation session.
  Evaluate the person's confidence in his or her balance, in the activities of daily living Simplified version of the "Activities-specific Balance Confidence scale between ¬60 to 70 days: the 20th and last rehabilitation session.
  Questionnaire made of 15 statements to assess the person's degree of confidence in his or her balance associated with activities of daily life in both the home environment and in the community environment. The questionnaire is part of this research administered by the evaluator.
  Add the scores obtained to the 15 items to obtain an overall score out of 45. The score is converted to a pourcentage.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte PANIGOT GUERIN, PT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Physique et de Réadaptation (MPR), Paris, France

REFERENCES:
- [Background] Barrois RP, Ricard D, Oudre L, Tlili L, Provost C, Vienne A, Vidal PP, Buffat S, Yelnik AP. Observational Study of 180 degrees Turning Strategies Using Inertial Measurement Units and Fall Risk in Poststroke Hemiparetic Patients. Front Neurol. 2017 May 15;8:194. doi: 10.3389/fneur.2017.00194. eCollection 2017. PMID 28555124
- [Background] Bonan IV, Yelnik AP, Colle FM, Michaud C, Normand E, Panigot B, Roth P, Guichard JP, Vicaut E. Reliance on visual information after stroke. Part II: Effectiveness of a balance rehabilitation program with visual cue deprivation after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2004 Feb;85(2):274-8. doi: 10.1016/j.apmr.2003.06.016. PMID 14966713
- [Background] Yelnik AP, Le Breton F, Colle FM, Bonan IV, Hugeron C, Egal V, Lebomin E, Regnaux JP, Perennou D, Vicaut E. Rehabilitation of balance after stroke with multisensorial training: a single-blind randomized controlled study. Neurorehabil Neural Repair. 2008 Sep-Oct;22(5):468-76. doi: 10.1177/1545968308315996. PMID 18780882
- [Background] Provost CP, Tasseel-Ponche S, Lozeron P, Piccinini G, Quintaine V, Arnulf B, Kubis N, Yelnik AP. Standing postural reaction to visual and proprioceptive stimulation in chronic acquired demyelinating polyneuropathy. J Rehabil Med. 2018 Feb 28;50(3):278-284. doi: 10.2340/16501977-2314. PMID 29313871
- [Background] Missaoui B, Thoumie P. Balance training in ataxic neuropathies. Effects on balance and gait parameters. Gait Posture. 2013 Jul;38(3):471-6. doi: 10.1016/j.gaitpost.2013.01.017. Epub 2013 Mar 5. PMID 23465318
- [Background] Filiatrault J, Gauvin L, Fournier M, Parisien M, Robitaille Y, Laforest S, Corriveau H, Richard L. Evidence of the psychometric qualities of a simplified version of the Activities-specific Balance Confidence scale for community-dwelling seniors. Arch Phys Med Rehabil. 2007 May;88(5):664-72. doi: 10.1016/j.apmr.2007.02.003. PMID 17466738